CLINICAL TRIAL: NCT00720538
Title: Randomized Controlled Double-blind Vs. Placebo Multicentre Study on the Safety and Effectiveness of Thalidomide in the Treatment of Refractory Crohn's Disease and Ulcerative Colitis.
Brief Title: Thalidomide in Pediatric Inflammatory Bowel Diseases.
Acronym: TALIBDP
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: IRCCS Burlo Garofolo (Other)
Collaborators: Ospedale Meyer (Other); Pediatric Gastroenterology Unit, IRCCS Gaslini, Genoa. (Unknown); Vittore Buzzi Children's Hospital (Other); University of Pisa (Other); University of Messina (Other); Università degli Studi di Brescia (Other); University of Trieste (Other)
Responsible Party: Principal Investigator, Alessandro Ventura, MD, IRCCS Burlo Garofolo
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TAL-005414-20
Record Dates: First submitted 2008-07-18; First posted 2008-07-22 (Estimated); Last update posted 2012-10-26 (Estimated); Status verified 2012-10

CONDITIONS: Inflammatory Bowel Diseases; Crohn's Disease; Ulcerative Colitis
Keywords: Inflammatory bowel diseases.; Crohn disease.; Ulcerative, colitis.; Randomised controlled trial.; Therapy.; Thalidomide.; Children.
MeSH Terms: conditions — Inflammatory Bowel Diseases; Crohn Disease; Colitis, Ulcerative | interventions — Thalidomide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Thalidomide
  Interventions: Drug: Thalidomide
- 2 (Placebo Comparator): Placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Thalidomide — Thalidomide 1.5-2.5 mg/kg/die once a day, at evening.
  Other Names: Thalidomide PHARMION; Thalidomid CELGENE
  Arms: 1
Drug: placebo — placebo capsules
  Arms: 2

SUMMARY:
Several open-label studies reported thalidomide efficacy in inducing clinical remission and steroid tapering in refractory Inflammatory Bowel diseases (IBD), both in adults and in children.

This is a randomized placebo controlled (RCT) double blind study, to evaluate the efficacy of thalidomide in inducing clinical remission at 8 weeks in refractory IBD patients aged 2-20 years.

The primary hypotheses of the study is that thalidomide would be more effective than placebo in inducing clinical remission.

The RCT phase is followed by a open-label phase, to further evaluate efficacy and safety of thalidomide in thalidomide responders, with a total follow up of one year.

DETAILED DESCRIPTION:
Inflammatory bowel diseases (IBD) are particularly debilitating. They present chronic-recurrent symptoms which often seriously affects the patient's quality of life, acute complications which may need surgical interventions and long-term risks as evolution in cancer for ulcerative colitis.

Although onset is most common in the third decade of life, more than one third of IBD cases are diagnosed before age sixteen, and these younger patients, especially with Crohn's disease, are increasing in Western countries. Recent studies in the United Kingdom, Sweden and the United States report an incidence of 5-7 new cases of IBD every year per 100,000 subjects < 16 years of age, with an increasing trend over the last two decades.

IBD-related morbidity causes special concern in childhood-onset cases, since the disease can compromise height and weight development. This is even worsened in patients with poor disease control, which need steroid treatment in multiple courses and/or for a long period of time.

There are various drugs and treatments available for the management of IBD, but some patients, during the course of the illness, become resistant to conventional treatment, or develop serious adverse effects to immunosuppressive drugs.

A particular challenge is represented by those patients (especially children) who fail to respond to conventional treatment, or are steroid-dependent, or suffer from serious side effects from steroids use.

Thalidomide was first marketed in the early 1960s as a sedative drug and sadly gained notoriety because of its teratogenic effect. After few years from this tragedy, thalidomide was rediscovered both as an immunomodulator and as an anti-inflammatory drug, with anti tumor necrosis factor-alfa properties.

Thalidomide is now approved for the treatment of multiple myeloma and erythema nodosum leprorum. It has also been tested, with beneficial effects, in a variety of inflammatory diseases, especially those involving the skin and mucous membranes: recurrent aphthous stomatitis, oral and oesophageal ulcers in HIV, oral and genital ulcers and intestinal symptoms in Behcet's syndrome, graft versus host disease, skin manifestations in systemic lupus erythematosus, sarcoidosis, and tuberculosis. In these diseases, especially in those cases resistant to conventional treatments, thalidomide seems to have a promising role as a secondary therapeutic option.

The safety and efficacy of thalidomide in IBD has been recently evaluated in several open-label studies both adults and children, some of which with a long-term follow up. A total of approximately 200 patients with steroid-resistant or steroid-dependent IBD were treated with thalidomide. Overall, the drug was effective in inducing clinical remission in 20-70% of patients (average of 40%). 60-100% patients (average of 70%) had some clinical response. Steroid-tapering was possible in 60-100% of cases.

The most frequent side effect of thalidomide in IBD cases was neuropathy, which mainly reported as cumulative dose-dependent. Other possible side effects are constipation, sedation, dermatitis, mood disturbance, vertigo, cephalea, hypertension, hormonal alterations.

In the experience of our center, thalidomide was effective in achieving clinical remission in several children, adolescents, and young adults with intractable IBD. From 1998 to 2004 twenty-eight patients with refractory moderate-severe IBD (19 CD, 9 UC) received thalidomide 1.5-2.5 mg/kg/day. Remission was achieved with thalidomide in 21 of 28 (75%) patients (17 with CD, 4 with UC). Mean duration of remission was 34.5 months. Sixteen of 20 (80%) patients suspended steroids. Reversible neuropathy occurred in seven of 28 (25%) patients, but only with cumulative doses over 28 g. Other side effects requiring thalidomide suspension were vertigo/somnolence (one case), and agitation/ hallucinations (one case).

The aim of this study is to evaluate the efficacy of thalidomide therapy in children, adolescents and young adults with refractory Crohn's disease (CD) and ulcerative colitis (UD), with a total follow up of one year.

The study is divided in two phases:

* Phase I: randomized placebo controlled double blind study, to evaluate efficacy of thalidomide in refractory IBD patients, at 8 weeks.
* Phase II: open-label study, to evaluate efficacy and safety of thalidomide in patients responders to Thalidomide in Phase I, with a total follow up of one year.

Analysis will be stratified for Crohn's disease and ulcerative colitis. Given the hypotheses that thalidomide will be effective in inducing clinical remission at 8 weeks in 60% of patients with Crohn's disease, and 55% of patients with ulcerative colitis, compared to 20% of patients with placebo, with a significance of 0.05% and a power of 80%, estimated needed sample size is of 124 patients.

ELIGIBILITY:
Inclusion Criteria:

* Children, adolescents and young adults aged 2 to 20 with chronic refractory moderate to severe inflammatory bowel disease, referred by the six pediatric gastroenterological centres participating in the study.

Definition of patient with refractory disease:

* Patients with active disease despite steroid therapy (prednisone at a dose 2 mg/kg/die, maximum 60mg/day, or equivalent) for 8 weeks and/or an immunosuppressive of proven efficacy (azathioprine o 6-mercaptopurine for 4 months; methotrexate for 3 months; Infliximab at the dose of 5 mg/kg at week 0,2,6 weeks; cyclosporine at the dose of 2mg/kg/day for 4 weeks or 1 week at 1m/kg/day EV) or patients exhibiting intolerance to these drugs which prevent them from continuing treatment.

Exclusion Criteria:

* Patients with ileostomy or colostomy.
* Disease requiring immediate surgical intervention.
* Severe ulcerative colitis or toxic megacolon.
* Contraindications to using thalidomide (on-going pregnancy, neuropathy) .
* Any of the following conditions: active infection, stool culture positive for enteric pathogens, tumors, HIV, transplanted organ, or non-controlled disease of the kidney, liver, endocrine system, heart, blood, nervous system or brain.
* Patients being treated with other drugs as part of an experimental study.
* Patients treated with infliximab in the previous eight weeks.

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 84 (Actual)
Dates: Start 2008-08; Primary Completion 2011-09 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Clinical Remission | 8°, 12°, 26, 52° weeks

SECONDARY OUTCOMES:
Clinical response | 4°, 8° weeks
Steroid dose reduction | 8°, 12°, 26, 52° weeks
Endoscopic remission | 12°, 26, 52° weeks
Adverse effects | 4°, 8°, 12°, 26, 52° weeks
Nutritinal indicators | 8°, 52°
  Weight-on-age z-scores (WAZ) 8°, 52° Body Mass Index (BMI) z-scores 8°, 52° Height-on-age z-scores (HAZ) 52°

CONTACTS AND LOCATIONS:
Overall Officials: Alessandro Ventura, MD, Study Chair — IRCCS Burlo Garofolo; Marzia Lazzerini, MD, Study Director — IRCCS Burlo Garofolo
Locations (7):
- Italy (7):
  - Anatomy and Hystology, Spedali Civili di Brescia, University of Brescia., Brescia, Brescia
  - Department of Pediatrics, Ospedale Meyer., Florence, Florence
  - Pediatric Gastroenterology Unit, IRCCS Gaslini., Genoa, Genoa
  - Pediatric Gastroenterology Unit, University of Messina., Messina, Messina
  - Department of Pediatrics, Ospedali Buzzi., Milan, Milan.
  - Gastroenterology and Hepatology, University of Pisa., Pisa, Pisa
  - Unit of Biochemistry and Pharmacology, University of Triest., Trieste, Triest

REFERENCES:
- [Background] Lazzerini M, Martelossi S, Marchetti F, Scabar A, Bradaschia F, Ronfani L, Ventura A. Efficacy and safety of thalidomide in children and young adults with intractable inflammatory bowel disease: long-term results. Aliment Pharmacol Ther. 2007 Feb 15;25(4):419-27. doi: 10.1111/j.1365-2036.2006.03211.x. PMID 17269997
- [Derived] Lazzerini M, Martelossi S, Magazzu G, Pellegrino S, Lucanto MC, Barabino A, Calvi A, Arrigo S, Lionetti P, Lorusso M, Mangiantini F, Fontana M, Zuin G, Palla G, Maggiore G, Bramuzzo M, Pellegrin MC, Maschio M, Villanacci V, Manenti S, Decorti G, De Iudicibus S, Paparazzo R, Montico M, Ventura A. Effect of thalidomide on clinical remission in children and adolescents with refractory Crohn disease: a randomized clinical trial. JAMA. 2013 Nov 27;310(20):2164-73. doi: 10.1001/jama.2013.280777. PMID 24281461